CLINICAL TRIAL: NCT01068509
Title: A Randomized, Open-label Phase IIb Trial of Maintenance Therapy With a MUC1 Dendritic Cell Vaccine (Cvac™) for Epithelial Ovarian Cancer Patients in First or Second Remission
Brief Title: Ovarian Cancer Vaccine for Patients in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prima BioMed Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN-003
Record Dates: First submitted 2010-02-10; First posted 2010-02-15 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2016-06

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Cvac
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — CCV-AV protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Non-randomized Cvac (Experimental): Participants received 6-8 intradermal injections of Cvac at 4 sites along both upper arms and both thighs. The 6-8 injections contained ~ 60 × 10^6 dendritic cells. Following evaluation after the first dose, participants received additional injections as described for the randomized Cvac group below.
  Interventions: Biological: Cvac
- Randomized Cvac (Experimental): Participants received 6-8 intradermal injections of Cvac at 4 sites along both upper arms and both thighs every 4 weeks for 24 weeks (7 doses at Weeks 8, 12, 16, 20, 24, 28, and 32), and then every 8 weeks for 24 weeks (3 doses at Weeks 40, 48, and 56). The 6-8 injections contained ~ 60 × 10^6 dendritic cells.
  Interventions: Biological: Cvac
- Observational standard of care (No Intervention): Participants in this group did not receive any treatment during the study.

INTERVENTIONS:
Biological: Cvac — Cvac consists of autologous dendritic cells (DCs) incubated with the antigen, mannosylated fusion protein (M-FP), to target the DCs to the specific mucin 1 antigen.
  Arms: Non-randomized Cvac; Randomized Cvac

SUMMARY:
The purpose of this study is to determine the safety and efficacy of an investigational therapeutic agent (Cvac) in ovarian cancer patients in first or second remission and to determine its ability to prevent cancer from returning.

Study objectives

Primary objectives:

* To confirm the safety of administering Cvac in this population.
* To determine the effects of Cvac on progression-free survival (PFS).

Secondary objectives:

* To determine overall survival (OS) for ovarian cancer patients who receive Cvac after achieving remission in the first or second-line setting.
* Evaluation of host immunologic response to Cvac administration.

DETAILED DESCRIPTION:
An initial cohort of 7 patients were treated with Cvac in an open-label phase to confirm the safety and consistency of manufacturing between Cvac drug product manufactured in the United States (US) and Australia. After the manufacturing characteristics of Cvac were confirmed to be consistent and each patient in the initial cohort had completed 1 injection cycle of Cvac with no serious or treatment-related Grade 3 or 4 adverse events (AEs), 56 patients were enrolled and randomized (1:1) to either Cvac or observational standard of care (OSC).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ≥ 18 years old with histologically confirmed Stage III or IV epithelial ovarian, primary peritoneal or fallopian tube cancer who have previously undergone surgical cytoreduction and received first or second line conventional chemotherapy and are currently in complete remission (based on clinical and radiologic studies).
* Cancer antigen (CA)-125 ≤ upper limit of normal with a prior history of an elevated CA-125.
* Able and willing to undergo mononuclear cell collection.
* Not more than 12 weeks between enrollment and the last dose of chemotherapy that resulted in complete remission.
* No prior surgery to the peritoneum or pleural space within 28 days of enrollment, excluding removal of catheters used for chemotherapy administration.
* No prior treatment with an investigational product within 30 days of enrollment.
* Baseline electrocardiogram within normal limits or any abnormalities deemed not indicative of cardiac disease for which intervention is required.
* Serum creatinine ≤ 2 mg/dL.
* Serum aspartate aminotransferase or serum alanine aminotransferase ≤ 2.5x the upper limit of normal or serum total bilirubin ≤ 1.5x the upper limit of normal.
* White blood cell count ≥ 3.0 K/µL; absolute neutrophil count ≥ 1.5K/µL; hemoglobin ≥ 9.0 g/dL, and platelets ≥ 100,000/mm^3. (These complete blood count results are required for enrollment. It should be noted that complete blood count results, including monocyte count ≥ 0.2 × 10^9/L, will be needed prior to leukapheresis to determine if sufficient dendritic cells can be obtained for Cvac™ manufacture.)
* Life expectancy of at least 12 months.
* Eastern Cooperative Oncology Group Performance Status of 0-1.
* All toxicities from prior therapies, excluding alopecia, must have resolved to Common Terminology Criteria for Adverse Events Grade ≤ 1.
* Must be non-pregnant and, if of childbearing potential, must use adequate birth control (hormonal or barrier method of birth control or abstinence) for the duration of the study and for 3 months after study completion.
* Able to provide written informed consent.

Exclusion Criteria:

* Coexisting or other malignancies unless in complete remission for not less than 3 years. Does not include in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin for which no restrictions apply, assuming they have been adequately treated.
* Ovarian germ cell, sarcoma, or mixed Mullerian tumors.
* Prior cancer vaccine or cellular therapy.
* Active uncontrolled infections or any organ system toxicity ≥ Grade 2 by Common Terminology Criteria for Adverse Events criteria.
* Inability to provide informed consent or to comply with study-related procedures.
* Concurrent systemic treatment with steroids or other immunosuppressive agents.
* Diagnosed immunodeficiency and/or autoimmune disorders.
* Myocardial infarction in the past 6 months and/or clinically significant heart disease.
* Infection with human immunodeficient virus (HIV), hepatitis B or C virus.
* Pregnant or breastfeeding.
* Evidence or history of central nervous system metastases.
* Full dose anticoagulation therapy administered within 7 days of leukapheresis procedure.
* Hematopoietic growth factors administered within 14 days of enrollment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Gray, MD, Principal Investigator — University of Washington; Mark Moradi, MD, Principal Investigator — New York Presbyterian Hospital; Jonathan Berek, MD, MMS, Principal Investigator — Stanford University; Nana Tchabo, MD, Principal Investigator — Morristown Medical Center; Jennifer Young, MD, Principal Investigator — Medical University of South Carolina; James Mason, MD, Principal Investigator — Scripps Cancer Center; Angeles Secord, MD, Principal Investigator — Duke University; Peter Eisenberg, MD, Principal Investigator — Marin Cancer Care; Giuseppe Del Priore, MD, Principal Investigator — Indiana University School of Medicine; Peter Rose, MD, Principal Investigator — The Cleveland Clinic; Fernando Recio, MD, Principal Investigator — Collaborative Research Group; Benedict Benigno, MD, Principal Investigator — Northside Hospital; John Chan, MD, Principal Investigator — University of California, San Francisco; Paul Mitchell, MB ChB, Principal Investigator — Austin Health Cancer Care; Linda Mileshkin, MBBS, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Margaret Davy, MBBS, CGO, Principal Investigator — Royal Adelaide Hospital; Jeffrey Goh, MBBS, FRACP, Principal Investigator — Greenslopes Private Hospital; Marco Matos, FRACP, Principal Investigator — Gold Coast Hospital
Locations (18):
- United States (13):
  - Marin Cancer Care, Inc., Greenbrae, California
  - Scripps Cancer Center, La Jolla, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Collaborative Research Group, Boca Raton, Florida
  - Northside Hospital, Atlanta, Georgia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Morristown Medical Center, Morristown, New Jersey
  - New York Downtown Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Washington Medical Center, Seattle, Washington
- Australia (5):
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Cetnre, East Melbourne, Victoria
  - Austin Health Cancer Centre, Heidelberg, Victoria

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Grossi M, Quinn MA, Thursfield VJ, Francis PA, Rome RM, Planner RS, Giles GG. Ovarian cancer: patterns of care in Victoria during 1993-1995. Med J Aust. 2002 Jul 1;177(1):11-6. doi: 10.5694/j.1326-5377.2002.tb04616.x. PMID 12088472
- [Background] Ozols RF, Rubin SC, Thomas G, et al. Epithelial ovarian cancer. In: Hoskins WJ, Perez CA, Young RC, eds. Principles and Practice of Gynecologic Oncology, 4th ed. Philadelphia: Lippincott Williams & Wilkins. 2005:919-922.
- [Background] Markman M, Liu PY, Wilczynski S, Monk B, Copeland LJ, Alvarez RD, Jiang C, Alberts D; Southwest Oncology Group; Gynecologic Oncology Group. Phase III randomized trial of 12 versus 3 months of maintenance paclitaxel in patients with advanced ovarian cancer after complete response to platinum and paclitaxel-based chemotherapy: a Southwest Oncology Group and Gynecologic Oncology Group trial. J Clin Oncol. 2003 Jul 1;21(13):2460-5. doi: 10.1200/JCO.2003.07.013. PMID 12829663
- [Background] Apostolopoulos V, McKenzie IF. Cellular mucins: targets for immunotherapy. Crit Rev Immunol. 1994;14(3-4):293-309. doi: 10.1615/critrevimmunol.v14.i3-4.40. PMID 7538768
- [Background] Desai J, Mitchell P, Loveland B, et al. A phase I trial of dendritic cells pulsed with MUC1 peptide in patients with solid tumours. Proc ASCO 2002; 21:15b (A1868).
- [Background] Rustin GJ, Nelstrop AE, Bentzen SM, Bond SJ, McClean P. Selection of active drugs for ovarian cancer based on CA-125 and standard response rates in phase II trials. J Clin Oncol. 2000 Apr;18(8):1733-9. doi: 10.1200/JCO.2000.18.8.1733. PMID 10764434
- [Background] Apostolopoulos V, McKenzie IF, Pietersz GA. Breast cancer immunotherapy: current status and future prospects. Immunol Cell Biol. 1996 Oct;74(5):457-64. doi: 10.1038/icb.1996.76. PMID 8912009
- [Background] Apostolopoulos V, Karanikas V, Haurum JS, McKenzie IF. Induction of HLA-A2-restricted CTLs to the mucin 1 human breast cancer antigen. J Immunol. 1997 Dec 1;159(11):5211-8. PMID 9548459
- [Background] Meyer T, Rustin GJ. Role of tumour markers in monitoring epithelial ovarian cancer. Br J Cancer. 2000 May;82(9):1535-8. doi: 10.1054/bjoc.2000.1174. PMID 10789720
- [Background] Liu PY, Alberts DS, Monk BJ, Brady M, Moon J, Markman M. An early signal of CA-125 progression for ovarian cancer patients receiving maintenance treatment after complete clinical response to primary therapy. J Clin Oncol. 2007 Aug 20;25(24):3615-20. doi: 10.1200/JCO.2006.09.4540. PMID 17704410
- [Background] Clinical Study Report: A Phase II Trial of Cellular Immunotherapy with M-FP Cancer Vaccine in Subjects with Epithelial Ovarian Cancer, 2007 (with permission from Martin Rogers of Prima Biomed).
- [Background] Immunotherapy for Prostate AdenoCarcinoma Treatment (IMPACT) Phase 3 study summary of sipuleucel-T in castrate-resistant prostate cancer: http://www.bio-medicine.org/medicine-technology-1/
- [Background] Austin Research Institute. SOP #811609. Leukapheresis for ex vivo Culture or Human Dendritic Cells for Immunotherapy. V004, 9 January 2004.
- [Background] Austin Research Institute. SOP #8116 Stages 3-4. Procedures for the ex vivo Generation of MF-P Vaccine Pulsed SC, Phase I Clinical Trial. V006, 10 June 2003.
- [Derived] Gray HJ, Benigno B, Berek J, Chang J, Mason J, Mileshkin L, Mitchell P, Moradi M, Recio FO, Michener CM, Secord AA, Tchabo NE, Chan JK, Young J, Kohrt H, Gargosky SE, Goh JC. Progression-free and overall survival in ovarian cancer patients treated with CVac, a mucin 1 dendritic cell therapy in a randomized phase 2 trial. J Immunother Cancer. 2016 Jun 21;4:34. doi: 10.1186/s40425-016-0137-x. eCollection 2016. PMID 27330807
- See also: Related Info from Sponsor's Web Site — http://primabiomed.com.au/investor/presentations.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-randomized Cvac | Randomized Cvac | Observational Standard of Care
Started | 7 | 29 | 27
Completed | 1 | 7 | 6
Not Completed | 6 | 22 | 21
Not completed — Death | 0 | 0 | 1
Not completed — Disease Progression | 5 | 20 | 18
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrew Consent | 0 | 1 | 2
Not completed — Reason Not Specified | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants: All participants enrolled in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-randomized Cvac | Randomized Cvac | Observational Standard of Care | Total
Number analyzed (Participants) | 7 | 29 | 27 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.4 (10.3) | 56.8 (8.5) | 56.2 (9.5) | 56.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 29 | 27 | 63
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the date of documented disease progression or death from any cause, whichever occurred earlier. Disease progression occurred when a patient met either the Gynecologic Cancer Intergroup (GCIG) cancer-antigen (CA)-125 definition or the Response Evaluation Criteria in Solid Tumors (RECIST) radiological definition of progressive disease. The GCIG CA-125 definition of disease progression was defined as a CA-125 level ≥ 2 × the upper limit of normal documented on 2 occasions at least 1 week apart. The radiological RECIST criteria of disease progression was defined as the appearance of new lesions or an overall increase ≥ 20% or at least 5 mm in existing tumors.
Time Frame: Baseline to 48 weeks after the last visit or dose of Cvac (up to 104 weeks)
Population: Intent-to-treat population: All randomized participants. Efficacy data were not collected on the initial cohort of 7 non-randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Cvac | Observational Standard of Care
Number analyzed (Participants) | 29 | 27
Months | 12.89 [7.26 to 22.77] | 8.64 [4.66 to 18.33]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause.
Time Frame: Baseline to the end of the study (up to 4 years 10 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized Cvac | Observational Standard of Care
Number analyzed (Participants) | 29 | 27
Months | NA [NA to NA] — The median (95% Confidence Interval) could not be calculated due to too few deaths. | NA [NA to NA] — The median (95% Confidence Interval) could not be calculated due to too few deaths.

3. Secondary Outcome: Change From Baseline in Mucin 1 Antibody Levels at Weeks 20, 56, and 104
Description: Mucin 1 antibodies were assessed in serum samples using a quantitative enzyme-linked immunosorbent assay (ELISA). Detection was achieved with electrochemiluminescence.
Time Frame: Baseline to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Randomized Cvac | Observational Standard of Care
Number analyzed (Participants) | 29 | 27
Arbitrary units
  Week 20 (n's=21, 13) | 957.2 (9127.3) | -2854.8 (9411.8)
  Week 56 (n's=8, 6) | -1113.9 (12033.3) | -19063.1 (41323.7)
  Week 104 (n's=10, 10) | -203.0 (4413.4) | -1956.7 (5711.1)

4. Secondary Outcome: Change From Baseline in ICS of IL2, IL4, IL17, TNF, and IFNg in CD4+ and CD8+ Cells at Weeks 20, 56, and 104
Description: Intracellular cytokine staining (ICS) for IL2, IL4, IL17, tumor necrosis factor (TNF), and interferon gamma (IFNg) was done in both CD4+ and CD8+ cells from serum samples collected at Weeks, 20, 56, and 104. Intracellular cytokine staining data were acquired with 8-color flow cytometry on a BD LSR II flow cytometer and a high-throughput screening microplate reader.
Time Frame: Baseline to Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Randomized Cvac | Observational Standard of Care
Number analyzed (Participants) | 29 | 27
Arbitrary units
  Week 20: IL2 in CD4+ cells (n's=21, 14) | -1.4022 (0.9730) | -1.1842 (1.0945)
  Week 20: IL4 in CD4+ cells (n's=21, 14) | -0.0702 (0.3781) | -0.1651 (0.2876)
  Week 20: IL17 in CD4+ cells (n's=21, 14) | -1.0544 (1.1481) | -0.3960 (0.4052)
  Week 20: TNF in CD4+ cells (n's=21, 14) | -2.7106 (2.1428) | -1.8939 (1.7481)
  Week 20: IFNg in CD4+ cells (n's=21, 14) | -1.3576 (1.5922) | -1.0243 (1.2047)
  Week 20: IL2 in CD8+ cells (n's=21, 14) | -0.3724 (0.3808) | -0.4562 (0.5527)
  Week 20: IL4 in CD8+ cells (n's=21, 14) | -0.1495 (0.1218) | -0.5607 (1.4552)
  Week 20: IL17 in CD8+ cells (n's=21, 14) | -0.8268 (1.6737) | -0.1232 (0.1367)
  Week 20: TNF in CD8+ cells (n's=21, 14) | -2.0802 (2.0004) | -1.9156 (2.1254)
  Week 20: IFNg in CD8+ cells (n's=21, 14) | -2.8385 (2.5259) | -2.3178 (2.1022)
  Week 56: IL2 in CD4+ cells (n's=2, 2) | -1.6798 (2.1394) | -1.6798 (2.1394)
  Week 56: IL4 in CD4+ cells (n's=2, 2) | -0.3824 (0.1417) | -0.3824 (0.1417)
  Week 56: IL17 in CD4+ cells (n's=2, 2) | -0.9413 (0.6249) | -0.9413 (0.6249)
  Week 56: TNF in CD4+ cells (n's=2, 2) | -5.9500 (3.3064) | -5.9500 (3.3064)
  Week 56: IFNg in CD4+ cells (n's=2, 2) | -1.2676 (0.4039) | -1.2676 (0.4039)
  Week 56: IL2 in CD8+ cells (n's=2, 2) | -0.9438 (0.0057) | -0.9438 (0.0057)
  Week 56: IL4 in CD8+ cells (n's=2, 2) | 0.0622 (0.0950) | -0.0622 (0.0950)
  Week 56: IL17 in CD8+ cells (n's=2, 2) | -0.0396 (0.0136) | -0.0396 (0.0136)
  Week 56: TNF in CD8+ cells (n's=2, 2) | -5.8027 (3.2811) | -5.8027 (3.2811)
  Week 56: IFNg in CD8+ cells (n's=2, 2) | -5.9300 (3.7024) | -5.9300 (3.7024)
  Week 104: IL2 in CD4+ cells (n's=3, 1) | -2.3179 (1.8772) | -1.4545 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IL4 in CD4+ cells (n's=3, 1) | -0.3328 (0.1972) | -0.2912 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IL17 in CD4+ cells (n's=3, 1) | -1.1783 (0.5970) | -1.0044 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: TNF in CD4+ cells (n's=3, 1) | -6.4140 (2.3691) | -2.9642 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IFNg in CD4+ cells (n's=3, 1) | -1.3833 (0.3474) | -1.5452 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IL2 in CD8+ cells (n's=3, 1) | -1.1586 (0.3643) | -0.1277 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IL4 in CD8+ cells (n's=3, 1) | -0.1241 (0.0688) | -0.1282 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IL17 in CD8+ cells (n's=3, 1) | -0.2485 (0.3395) | -0.4682 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: TNF in CD8+ cells (n's=3, 1) | -5.1697 (2.6055) | -1.6795 (NA) — The standard deviation could not be calculated as there was only 1 participant.
  Week 104: IFNg in CD8+ cells (n's=3, 1) | -5.1340 (3.0755) | -2.3506 (NA) — The standard deviation could not be calculated as there was only 1 participant.

ADVERSE EVENTS:
Description: Safety population: All participants who received at least 1 dose of Cvac or were assigned to the observational standard of care group and were assessed at Week 20 (7 participants in the initial cohort, 26 of 29 participants randomized to Cvac, and 24 of 27 participants randomized to observational standard of care).
Arm/Group | Non-randomized Cvac | Randomized Cvac | Observational Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/7 | 4/26 | 0/24
Other Adverse Events (participants affected / at risk) | 7/7 | 25/26 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized Cvac (N=7) | Randomized Cvac (N=26) | Observational Standard of Care (N=24)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Ovarian epithelial cancer metastatic (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-randomized Cvac (N=7) | Randomized Cvac (N=26) | Observational Standard of Care (N=24)
Fatigue (General disorders) | 1 | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 1 | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 6
Nausea (Gastrointestinal disorders) | 0 | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Urinary tract infection (Renal and urinary disorders) | 0 | 5 | 4
Constipation (Gastrointestinal disorders) | 0 | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Hot flush (Vascular disorders) | 1 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 4
Injection site erythema (Injury, poisoning and procedural complications) | 1 | 4 | 0
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Oedema peripheral (Metabolism and nutrition disorders) | 1 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 2
Injection site pain (Injury, poisoning and procedural complications) | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Pain (General disorders) | 0 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Depression (Psychiatric disorders) | 0 | 2 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 0 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Injection site reaction (Injury, poisoning and procedural complications) | 0 | 3 | 0
Lethargy (General disorders) | 0 | 2 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 2 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 2 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Renal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Vulvovaginal candidiasis (Reproductive system and breast disorders) | 0 | 2 | 0
Asthma (Immune system disorders) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Pelvic fluid collection (Gastrointestinal disorders) | 1 | 0 | 0
Right atrial dilatation (Cardiac disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For study centers in Australia, no publication of the study results may be made until publication of the results of the study from all centers or until 2 years after study completion, whichever is sooner. For study centers in the USA, no submission for publication or public disclosure of the results by will be made until the results from all centers have been received and analyzed by the sponsor, or the multi-center study has been terminated or abandoned at all centers.